CLINICAL TRIAL: NCT00524069
Title: A Pilot Study of Bevacizumab Based Peri-Operative Therapy for Operable Pancreatic Adenocarcinoma
Brief Title: Gemcitabine, Capecitabine, and Bevacizumab in Treating Patients With Pancreatic Cancer That Can Be Removed By Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to no accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: I 68805; RPCI-I-68805
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Capecitabine; Gemcitabine; Flow Cytometry; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: capecitabine
Drug: gemcitabine hydrochloride
Other: flow cytometry
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: computed tomography
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving gemcitabine and capecitabine together with bevacizumab may kill more tumor cells.

PURPOSE: This clinical trial is studying the side effects and how well giving gemcitabine and capecitabine together with bevacizumab works in treating patients with pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility and safety of bevacizumab-based neoadjuvant and adjuvant therapy in patients with resectable pancreatic adenocarcinoma.
* To determine the proportion of patients with margin-positive resections after pancreatic resection.

Secondary

* To estimate overall survival of patients treated with this regimen.
* To assess the time to recurrence in patients treated with this regimen.
* To measure the change in the number of circulating endothelial precursor cells (CEC) and VEGF expression on CEC at baseline and after the start of neoadjuvant therapy and examine their relationship with response, time to recurrence, and survival.
* To assess the utility of dynamic contrast-enhanced spiral CT scan as surrogate endpoints for antiangiogenic therapy.

OUTLINE: This is a multicenter study.

* Neoadjuvant therapy: Patients receive gemcitabine IV over 30 minutes on days 1 and 8; oral capecitabine twice daily on days 1-14; and bevacizumab* IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receive bevacizumab during courses 1 and 2 only.

* Surgical resection: Within 6-8 weeks after the last dose of bevacizumab, patients undergo surgical resection of the pancreatic tumor.
* Adjuvant therapy: Beginning 6-10 weeks after surgery, patients receive up to 6 additional courses of gemcitabine, capecitabine, and bevacizumab as in neoadjuvant therapy.

Patients undergo blood sample collection at baseline and periodically during study for biomarker correlative studies. Samples are analyzed by flow cytometry to measure levels of circulating endothelial precursor cells and VEGF markers of angiogenesis. Patients also undergo dynamic contrast-enhanced (DCE) spiral CT scan of the abdomen. DCE-CT imaging studies are performed at baseline and after completion of neoadjuvant therapy (1-2 weeks prior to surgical resection) to assess changes in tumor blood flow, blood volume, and tumor vasculature.

After completion of study therapy, patients are followed periodically for at least 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Resectable disease (i.e., stage I or II disease)

    * No unresectable (i.e., locally advanced) disease
* No tumor invasion into the stomach or duodenum
* No CNS, brain, or systemic metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC > 3,000/μL
* ANC > 1,500/μL
* Platelet count > 100,000/μL
* Total bilirubin < 2 mg/dL
* AST or ALT < 2.5 times upper limit of normal (ULN)
* Creatinine < 1.5 mg/dL
* Creatinine clearance ≥ 50 mL/min
* Urine protein:creatinine ratio < 1.0
* Hemoglobin ≥ 9 g/dL (transfusion, epoetin alfa, or darbepoetin allowed)
* INR < 1.5 times ULN (except in patients receiving full-dose warfarin)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled hypertension
* No unstable angina
* No New York Heart Association class II-IV congestive heart failure
* No myocardial infarction or stroke within the past 6 months
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No esophageal or gastric varices
* No serious nonhealing wound, ulcer, or bone fracture

PRIOR CONCURRENT THERAPY:

* No prior therapy for pancreatic cancer
* More than 4 weeks since prior and no concurrent participation in another experimental drug study
* More than 28 days since prior major surgical procedure or open biopsy
* More than 7 days since prior minor surgical procedure (e.g., fine-needle aspiration or core biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety
Margin status after pancreatic resection

SECONDARY OUTCOMES:
Proportion of patients with positive resection margins, including microscopic (R1) or gross (R2) positive resection margins
Median survival
Time to recurrence
Overall survival
Number of circulating endothelial precursor cells (CEC) and their VEGFR expression as measured by flow cytometry at baseline and after the start of neoadjuvant therapy
Correlation of CEC number and VEGFR expression with margin positivity, survival, and recurrence
Changes in blood volume, blood flow, mean transit time, and color flow maps of the tumor as measured by dynamic contrast-enhanced spiral CT scan at baseline and after completion of neoadjuvant therapy
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institute